CLINICAL TRIAL: NCT06539182
Title: A Phase 2, Open-label, Multicenter Study to Evaluate the Efficacy, Safety, Tolerability and Pharmacokinetics of DZD8586 in Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Brief Title: DZD8586 in Patients With Relapsed or Refractory CLL/SLL (TAI-SHAN8)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dizal Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DZ2023B0002
Record Dates: First submitted 2024-08-01; First posted 2024-08-06 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Daily dose of DZD8586 at 25 mg (Experimental)
  Interventions: Drug: DZD8586
- Daily dose of DZD8586 at 50 mg (Experimental)
  Interventions: Drug: DZD8586
- Daily dose of DZD8586 at 75 mg (Experimental)
  Interventions: Drug: DZD8586

INTERVENTIONS:
Drug: DZD8586 — Daily oral dose of DZD8586 at 25 mg.
  Other Names: Birelentinib
  Arms: Daily dose of DZD8586 at 25 mg
Drug: DZD8586 — Daily oral dose of DZD8586 at 50 mg.
  Other Names: Birelentinib
  Arms: Daily dose of DZD8586 at 50 mg
Drug: DZD8586 — Daily oral dose of DZD8586 at 75 mg.
  Other Names: Birelentinib
  Arms: Daily dose of DZD8586 at 75 mg

SUMMARY:
This study will treat patients with CLL/SLL whose disease comes back or is not responding to prior therapy, or if they can not bear side effects of the prior treatment. This study will assess the anti-tumor activity of DZD8586 as monotherapy. It will help to understand what type of side effects may occur with the drug treatment. It will also measure the levels of drug in the body.

ELIGIBILITY:
Inclusion Criteria:

Participants who meet all the following criteria:

1. Male and female ≥ 18 years of age.
2. ECOG performance status 0-2.
3. Confirmed diagnosis of CLL/SLL with indication for treatment.
4. Adequate bone marrow reserve and organ system functions.
5. Willing to comply with contraceptive restrictions.

Exclusion Criteria:

Participants who meet any of the following criteria:

1. CNS involvement or Richter transformation.
2. Stem cell transplantation, cell therapy, or gene therapy within 90 days. Approved small molecule therapy within 5 half-lives, monoclonal antibodies and antibody-drug conjugates within 28 days.
3. Major surgery or significant traumatic injury within 4 weeks. Live attenuated vaccines or viral vector vaccines within 4 weeks.
4. Take vitamin K antagonists or take more than 2 anticoagulants or antiplatelet drugs at the same time. Take proton pump inhibitors or strong CYP3A inhibitors or inducers.
5. Active infection.
6. Clinically significant cardiac disorders or abnormalities. History of thrombotic diseases, stroke or intracranial hemorrhage within 6 months.
7. Nausea and vomiting not controlled or chronic gastrointestinal diseases, unable to swallow the formulated product or previous bowel resection that would preclude adequate absorption.
8. Another malignancy within 2 years prior to enrollment with the exception of adequately treated in-situ carcinoma of the cervix, uterus, basal or squamous cell carcinoma or non-melanomatous skin cancer.
9. Women who are breast feeding.
10. History of hypersensitivity to active or inactive excipients of DZD8586 or drugs with a similar chemical structure or class.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate assessed by investigators | assessed up to 2 years

SECONDARY OUTCOMES:
Incidence of adverse event | 30 days after the last dose, assessed up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jianyong Li, Principal Investigator — First Affiliated Hospital of Nanjing Medical University, Jiangsu Province Hospital
Locations (14):
- China (14):
  - Research Site, Hefei, Anhui
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Guangzhou, Guandong
  - Research Site, Zhengzhou, Henan
  - Research Site, Wuhan, Hubei
  - First Affiliated Hospital of Nanjing Medical University, Jiangsu Province Hospital, Nanjing, Jiangsu
  - Research Site, Changchun, Jilin
  - Research Site, Dalian, Liaoning
  - Research Site, Shenyang, Liaoning
  - Research Site, Jinan, Shandong
  - Research Site, Linyi, Shandong
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Taiyuan, Shangxi
  - Research Site, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No